CLINICAL TRIAL: NCT00824265
Title: A Phase III, Open Label, Randomized Trial of Ofatumumab Added to Fludarabine-Cyclophosphamide vs. Fludarabine-Cyclophosphamide Combination in Subjects With Relapsed Chronic Lymphocytic Leukemia
Brief Title: Ofatumumab Added to Fludarabine-Cyclophosphamide vs Fludarabine-Cyclophosphamide Combination in Relapsed Subjects With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110913
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: Relapsed; Oncology; Safety; Chronic Lymphocytic Leukemia; Ofatumumab; Efficacy
MeSH Terms: conditions — Leukemia, B-Cell; Recurrence; Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ofatumumab, Fludarabine, Cyclophosphamide (Experimental): Ofatumumab Cycle 1-Day 1 300mg, Cycle 1-Day 8 1000mg, then Cycles 2-6 Day 1 1000mg every 28 days, Fludarabine 25mg/m2 Days 1-3 every 28 days for 6 cycles, Cyclophosphamide 250 mg/m2 Days 1-3 every 28 days for 6 cycles
  Interventions: Drug: OFC Infusion
- Fludarabine, Cyclophosphamide (Active Comparator): Fludarabine 25mg/m2 Days 1-3 every 28 days for 6 cycles, Cyclophosphamide 250 mg/m2 Days 1-3 every 28 days for 6 cycles
  Interventions: Drug: FC infusion

INTERVENTIONS:
Drug: OFC Infusion — Ofatumumab Cycle 1-Day 1 300mg, Cycle 1-Day 8 1000mg, then Cycles 2-6 Day 1 1000mg every 28 days, Fludarabine 25mg/m2 Days 1-3 every 28 days for 6 cycles, Cyclophosphamide 250 mg/m2 Days 1-3 every 28 days for 6 cycles
  Arms: Ofatumumab, Fludarabine, Cyclophosphamide
Drug: FC infusion — Fludarabine 25mg/m2 Days 1-3 every 28 days for 6 cycles, Cyclophosphamide 250mg/m2 Days 1-3 every 28 days for 6 cycles
  Arms: Fludarabine, Cyclophosphamide

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ofatumumab added to fludarabine-cyclophosphamide in patients with relapsed Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
Fludarabine is currently approved for treatment of relapsed Chronic Lymphocytic Leukemia. Studies have shown that drugs in combination with fludarabine have shown more effectiveness than fludarabine alone. The addition of ofatumumab to fludarabine-cyclophosphamide combination offers potentially a more effective therapy, without additional toxicity.

The objective of this study was to determine the effect of ofatumumab added to fludarabine and cyclophosphamide in patients with Chronic Lymphocytic Leukemia who have responded previously to therapy but later develop progressive disease and require additional therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* confirmed and active CLL requiring treatment
* at least one previous treatment for CLL and having achieved a complete or partial remission/response but after a period of 6 or more months, shows evidence of disease progression
* fully active at a minimum or fully capable of selfcare and up and about more than 50% of waking hours
* age 18yrs or older
* signed written informed consent

Key Exclusion Criteria:

* diagnosis of refractory CLL (failure to achieve a complete or partial remission/response or disease progression within 6 months of last anti-CLL treatment
* abnormal/inadequate blood values, liver and kidney function
* certain heart problems, serious significant diseases, AIHA, other current cancers or within the last 5 years
* active or chronic infections
* use of drugs to suppress allergic or inflammatory responses (glucocorticoids)
* CLL transformation
* CLL central nervous system involvement
* current participation in other clinical study
* inability to comply with the protocol activities
* lactating or pregnant women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2009-03-12 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (112):
- United States (6):
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Clinton, Maryland
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Memphis, Tennessee
- Brazil (7):
  - Novartis Investigative Site, Brasilia, Goiás
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigational Site, Porto Alegre
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigation Site, Rio de Janeiro
  - Novartis Investigational Site, São Paulo
- Bulgaria (5):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigational Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (8):
  - Novartis Investigative Site, New Westminster, British Columbia
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Germany (15):
  - Novartis Investigative Site, Karlsruhe, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Villingen-Schwenningen, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Lehrte, Lower Saxony
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Moenchengladbach-Rheydt, North Rhine-Westphalia
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Saarbrücken, Saarland
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigational Site, Hamburg
  - Novartis Investigational Site, Lübeck
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- India (5):
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Pune
  - Novartis Investigative Site, Vadodara
- Italy (9):
  - Novartis Investigative Site, Potenza, Basilicate
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Pavia, Lombardy
  - Novartis Investigative Site, Alessandria, Piedmont
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Catania, Sicily
  - Novartis Investigative Site, Palermo, Sicily
  - Novartis Investigative Site, Ascoli Piceno, The Marches
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mexico City
- Netherlands (4):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, The Hague
- Poland (9):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Romania (3):
  - Novartis Investigative Site, Bucharest
  - Iași
  - Novartis Investigative Site, Iași
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
- Spain (4):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigational Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- Ukraine (10):
  - Novartis Investigative Site, Cherkasy
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Khmelnytskyi
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Makiivka
  - Novartis Investigational Site, Simferopil
  - Novartis Investigative Site, Vinnitsa
  - Novartis Investigational Site, Zhytomyr
- United Kingdom (13):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Burton-on-Trent
  - Novartis Investigative Site, Cottingham
  - Novartis Investigative Site, Dudley
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Sutton
  - Novartis Investigative Site, Swindon
  - Novartis Investigative Site, Truro
  - Novartis Investigative Site, Uxbridge

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Robak T, Warzocha K, Govind Babu K, Kulyaba Y, Kuliczkowski K, Abdulkadyrov K, Loscertales J, Kryachok I, Kloczko J, Rekhtman G, Homenda W, Blonski JZ, McKeown A, Chang CN, Bal V, Lisby S, Gupta IV, Grosicki S. Health-related quality of life and patient-reported outcomes of ofatumumab plus fludarabine and cyclophosphamide versus fludarabine and cyclophosphamide in the COMPLEMENT 2 trial of patients with relapsed CLL. Leuk Lymphoma. 2017 Jul;58(7):1598-1606. doi: 10.1080/10428194.2016.1253837. Epub 2016 Nov 10. PMID 27830957
- [Derived] Robak T, Warzocha K, Govind Babu K, Kulyaba Y, Kuliczkowski K, Abdulkadyrov K, Loscertales J, Kryachok I, Kloczko J, Rekhtman G, Homenda W, Blonski JZ, McKeown A, Gorczyca MM, Carey JL, Chang CN, Lisby S, Gupta IV, Grosicki S. Ofatumumab plus fludarabine and cyclophosphamide in relapsed chronic lymphocytic leukemia: results from the COMPLEMENT 2 trial. Leuk Lymphoma. 2017 May;58(5):1084-1093. doi: 10.1080/10428194.2016.1233536. Epub 2016 Oct 12. PMID 27731748
- [Derived] Jewell RC, Laubscher K, Lewis E, Fang L, Gafoor Z, Carey J, McKeown A, West S, Wright O, Sedoti D, Dixon I, Hottenstein CS, Chan G. Assessment of the effect of ofatumumab on cardiac repolarization. J Clin Pharmacol. 2015 Jan;55(1):114-21. doi: 10.1002/jcph.376. Epub 2014 Aug 21. PMID 25103870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par) were screened within 14 days prior to the start of study drug administration to determine eligibility.
Pre-assignment Details: Eligible par were stratified by Stage (Binet A vs. B vs. C) and number of prior therapies (1-2 vs. ≥3). Par in each stratum were then centrally randomized in a 1:1 ratio to recive intravenous (IV) fludarabine and cyclophosphamide in combination with ofatumumab or IV fludarabine and cyclophosphamide alone.
Groups:
- Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects: Participants with relapsed CLL received IV infusions of ofatumumab in combination with fludarabine and cyclophosphamide IV infusions for 6 cycles; each cycle comprised of 28 days. Participants received ofatumumab administered at 300 milligram (mg) on Day 1, 1000 mg on Day 8 of cycle 1 and 1000 mg on Day 1 of cycles 2, 3, 4, 5 and 6. Fludarabine was administered at 25 mg/meter squared [m^2] and cyclophosphamide was administered at 250mg/m^2 on Days 1-3 of each cycles (6 cycles). Participants were followed up one month post therapy and every 3 months for 5 years to evaluate survival and disease status.
- Fludarabine + Cyclophosphamide_ ITT Subjects: Participants with relapsed CLL received IV infusions of fludarabine administered at 25 mg/m^2 and cyclophosphamide administered at 250mg/m^2 on Days 1-3 of each cycle (6 cycles). Participants were followed up one month post therapy and every 3 months for 5 years to evaluate survival and disease status.
Period: Treatment Phase
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Started | 183 | 182
Completed | 119 | 102
Not Completed | 64 | 80
Not completed — Adverse Event,non-fatal | 50 | 52
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 6 | 12
Not completed — Withdrawal by Subject | 6 | 15
Period: Follow-up Phase
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Started | 172 | 160
Completed | 154 | 129
Not Completed | 18 | 31
Not completed — w/drew consent, no f/u, or MD choice | 18 | 31
Period: Survival Follow-up Phase
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Started | 96 | 89
Completed | 87 | 73
Not Completed | 9 | 16
Not completed — w/drew consent, no f/u, or MD choice | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects | Total
Number analyzed (Participants) | 183 | 182 | 365
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (8.82) | 61.6 (10.21) | 61.5 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 66 | 145
  Male | 104 | 116 | 220
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 3 | 5 | 8
  American Indian or Alaska Native | 3 | 1 | 4
  Asian - Central/South Asian Heritage | 13 | 16 | 29
  Asian - East Asian Heritage | 3 | 3 | 6
  Asian - South East Asian Heritage | 3 | 3 | 6
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 158 | 153 | 311

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS), as Assessed by the Independent Review Committee (IRC)
Description: PFS is defined as the interval of time between the date of randomization and the earlier of the date of disease progression (progressive disease,PD) and the date of death due to any cause. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlargerd lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia (CLL).
Time Frame: From randomization up to 5 years after last dose of study drug
Population: Intent-to-Treat (ITT) Population: all participants randomized and received study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Months | 28.94 [22.80 to 35.88] | 18.83 [14.42 to 25.82]
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.0032, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.51 to 0.88]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death due to any cause. Each participant was followed at the time when the last IRC-assessed PFS events occurred. Participants who had not died were censored at the date of last contact.
Time Frame: From randomization up to 5 years after last dose of study drug
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Months | 62.65 [44.58 to NA] — Upper limit was not able to calculate due to an insufficient number of events (high censoring rate) and high follow-up time | 46.23 [37.72 to 56.57]
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.1427, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.59 to 1.09]

3. Secondary Outcome: Time to Response, as Assessed by the IRC
Description: Time to response is defined as the time from randomization to the first response. Complete Response/remission(CR) all the criteria at least 2 months after last treatment: no lymphadenopathy(Ly) > 1.5 cm/ hepatomegaly/spleenomegaly/constitutional symptoms; neutrophils >1500 per microliter(µL), platelets(PL) >100,000/µL, hemoglobin(Hb) >11 grams/deciliter(g/dL), lymphocytes(LC) <4000/µL, bone marrow(BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. Incomplete bone marrow recovery(CRi): CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. Partial Remission/response(PR): >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline(BL), Hb >11 g/dL or 50% improvement over BL. Nodular PR(nPR): persistent nodules BM.
Time Frame: From randomization up to 5 years after last dose of study drug
Population: ITT Population. Participants with unknown or missing responses were considered as non-responders. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 152 | 123
Months | 0.99 [0.95 to 1.08] | 0.99 [0.95 to 1.18]
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.4490, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.85 to 1.37]

4. Secondary Outcome: Duration of Response (DOR), as Assessed by the IRC
Description: DOR is defined as the time from the initial response (CR, CRi, nPR, or PR) to the first documented sign of PD or death due to any cause. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlargerd lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia.
Time Frame: From time of initial response to disease progression or death, whichever came first (up to 5 years after the last dose of study drug)
Population: ITT Population. Par with unknown or missing responses were considered as non-responders, only responders were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 152 | 123
Months | 29.63 [25.03 to 41.46] | 24.90 [18.99 to 28.12]
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.0878, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.56 to 1.05]

5. Secondary Outcome: Time to Progression, as Assessed by the IRC
Description: Time to progression is defined as the time from the date of randomization to PD. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlargerd lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia.
Time Frame: From randomization up to 5 years after the last dose of study drug
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Months | 42.12 [28.94 to 47.67] | 26.78 [22.51 to 31.87]
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.0036, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.45 to 0.87]

6. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy is defined as the time from randomization until the start of the next-line of treatment. Data are presented for participants who took anti-cancer therapies and participants in the ITT population.
Time Frame: From the start of study drug until the start of the next anti-CLL therapy (up to 5 years after the last dose of study drug)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ofatumumab+Fludarabine+Cyclophosphamide_anti-CLL Therapies; Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects: Participants with relapsed CLL received IV infusions of ofatumumab in combination with fludarabine and cyclophosphamide IV infusions for 6 cycles; each cycle comprised of 28 days. Participants received ofatumumab administered at 300 milligram (mg) on Day 1, 1000 mg on Day 8 of cycle 1 and 1000 mg on Day 1 of cycles 2, 3, 4, 5 and 6. Fludarabine was administered at 25 mg/meter squared [m^2] and cyclophosphamide was administered at 250mg/m^2 on Days 1-3 of each cycles (6 cycles). Participants were followed up one month post therapy and every 3 months for 5 years to evaluate survival and disease status.
- Fludarabine+Cyclophosphamide_anti-CLL Therapies; Fludarabine + Cyclophosphamide_ ITT Subjects: Participants with relapsed CLL received IV infusions of fludarabine administered at 25 mg/m^2 and cyclophosphamide administered at 250mg/m^2 on Days 1-3 of each cycle (6 cycles). Participants were followed up one month post therapy and every 3 months for 5 years to evaluate survival and disease status.
Arm/Group | Ofatumumab+Fludarabine+Cyclophosphamide_anti-CLL Therapies | Fludarabine+Cyclophosphamide_anti-CLL Therapies | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 74 | 67 | 183 | 182
Months | 29.68 [24.97 to 32.66] | 21.03 [16.79 to 28.35] | 52.96 [43.56 to 62.98] | 40.08 [32.85 to 48.39]
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other — Participants in the ITT population; p = 0.1143, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.55 to 1.08]
Statistical Analysis 2: Comparison: Ofatumumab+Fludarabine+Cyclophosphamide_anti-CLL Therapies vs Fludarabine+Cyclophosphamide_anti-CLL Therapies; Test type: Superiority or Other — Participants who took anti-cancer therapies; p = 0.0109, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.48 to 0.94]

7. Secondary Outcome: Number of Participants With Improvement in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status scales and criteria are used by doctors and researchers to assess how a participant's disease is progressing, how the disease affects the daily living, and determines appropriate treatment and prognosis. ECOG performance status are measured at Cycle 2 Day1, Cycle 3 Day1, Cycle 4 Day1, Cycle 5 Day1 and Cycle 6 Day1. During follow period, 1 M after study drug therapy, then every 3 month up to 5 year (up to 60 months). Improvement is defined as a decrease from baseline by at least one step on the ECOG performance status scale (yes/no).
Time Frame: Cycle 2 Day1, Cycle 3 Day1, Cycle 4 Day1, Cycle 5 Day1, Cycle 6 Day1, follow up (FU) at 1Month (M) after study drug therapy, 3M, then every 3 month up to 5 year (up to 60 months)
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Participants
  Cycle 2 Day 1: number analyzed (Participants) | 170 | 168
  Cycle 2 Day 1 | 15 | 13
  Cycle 3 Day 1: number analyzed (Participants) | 165 | 157
  Cycle 3 Day 1 | 16 | 13
  Cycle 4 Day 1: number analyzed (Participants) | 153 | 132
  Cycle 4 Day 1 | 19 | 13
  Cycle 5 Day 1: number analyzed (Participants) | 135 | 118
  Cycle 5 Day 1 | 20 | 15
  Cycle 6 Day 1: number analyzed (Participants) | 120 | 96
  Cycle 6 Day 1 | 26 | 16
  1 M, FU: number analyzed (Participants) | 159 | 145
  1 M, FU | 31 | 22
  3 M, FU: number analyzed (Participants) | 152 | 119
  3 M, FU | 31 | 21
  6 M, FU: number analyzed (Participants) | 136 | 104
  6 M, FU | 30 | 18
  9 M, FU: number analyzed (Participants) | 127 | 96
  9 M, FU | 31 | 23
  12 M, FU: number analyzed (Participants) | 118 | 87
  12 M, FU | 30 | 20
  15 M, FU: number analyzed (Participants) | 102 | 70
  15 M, FU | 23 | 18
  18 M, FU: number analyzed (Participants) | 96 | 65
  18 M, FU | 23 | 18
  21 M, FU: number analyzed (Participants) | 92 | 59
  21 M, FU | 22 | 16
  24 M, FU: number analyzed (Participants) | 80 | 53
  24 M, FU | 20 | 15
  27 M, FU: number analyzed (Participants) | 74 | 44
  27 M, FU | 15 | 13
  30 M, FU: number analyzed (Participants) | 69 | 35
  30 M, FU | 14 | 8
  33 M, FU: number analyzed (Participants) | 65 | 29
  33 M, FU | 15 | 7
  36 M, FU: number analyzed (Participants) | 58 | 23
  36 M, FU | 12 | 7
  39 M, FU: number analyzed (Participants) | 51 | 18
  39 M, FU | 12 | 7
  42 M, FU: number analyzed (Participants) | 44 | 16
  42 M, FU | 11 | 6
  45 M, FU: number analyzed (Participants) | 39 | 14
  45 M, FU | 8 | 4
  48 M, FU: number analyzed (Participants) | 37 | 12
  48 M, FU | 8 | 2
  51 M, FU: number analyzed (Participants) | 32 | 12
  51 M, FU | 7 | 3
  54 M, FU: number analyzed (Participants) | 30 | 9
  54 M, FU | 7 | 2
  57 M, FU: number analyzed (Participants) | 26 | 9
  57 M, FU | 3 | 3
  60 M, FU: number analyzed (Participants) | 26 | 8
  60 M, FU | 3 | 3

8. Secondary Outcome: Number of Participants With no B-Symptoms or at Least One B-symptoms Over the Time
Description: Participants with no B-symptoms (B-Sy) (no night sweat, no weight loss, no fever and no extreme fatigue) and at least one indicated B-sy(night sweats, weight loss, fever or extreme fatigue) were presented at Screening, Cycle 1 Day 1, Cycle 2 Day1, Cycle 3 Day1, Cycle 4 Day1, Cycle 5 Day1, Cycle 6 Day 1 and during follow up period at 1 M after study drug therapy, then every 3 M up to 5 year (up to 60 months).
Time Frame: Screening, Cycle1 Day 1, Cycle 2 Day1, Cycle 3 Day1, Cycle 4 Day1, Cycle 5 Day1, Cycle 6 Day 1 and During at 1M after study drug therapy, 3M, then every 3 M up to 5 year (up to 60 months)
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Participants
  Screening, no B-sy: number analyzed (Participants) | 183 | 180
  Screening, no B-sy | 63 | 59
  Screening, one B-sy: number analyzed (Participants) | 183 | 180
  Screening, one B-sy | 120 | 121
  Cycle 1 Day 1, no B-sy: number analyzed (Participants) | 179 | 179
  Cycle 1 Day 1, no B-sy | 64 | 68
  Cycle 1 Day 1, one B-sy: number analyzed (Participants) | 179 | 179
  Cycle 1 Day 1, one B-sy | 115 | 111
  Cycle 2 Day 1,no B-sy: number analyzed (Participants) | 168 | 170
  Cycle 2 Day 1,no B-sy | 116 | 108
  Cycle 2 Day 1, one B-sy: number analyzed (Participants) | 168 | 170
  Cycle 2 Day 1, one B-sy | 52 | 62
  Cycle 3 Day 1, no B-sy: number analyzed (Participants) | 165 | 156
  Cycle 3 Day 1, no B-sy | 131 | 116
  Cycle 3 Day 1, one B-sy: number analyzed (Participants) | 165 | 156
  Cycle 3 Day 1, one B-sy | 34 | 40
  Cycle 4 Day 1, no B-sy: number analyzed (Participants) | 154 | 132
  Cycle 4 Day 1, no B-sy | 129 | 107
  Cycle 4 Day 1, one B-sy: number analyzed (Participants) | 154 | 132
  Cycle 4 Day 1, one B-sy | 25 | 25
  Cycle 5 Day 1, no B-sy: number analyzed (Participants) | 134 | 118
  Cycle 5 Day 1, no B-sy | 120 | 97
  Cycle 5 Day 1, one B-sy: number analyzed (Participants) | 134 | 118
  Cycle 5 Day 1, one B-sy | 14 | 21
  Cycle 6 Day 1, no B-sy: number analyzed (Participants) | 120 | 95
  Cycle 6 Day 1, no B-sy | 111 | 82
  Cycle 6 Day 1, one B-sy: number analyzed (Participants) | 120 | 95
  Cycle 6 Day 1, one B-sy | 9 | 13
  1 M, FU, no B-sy: number analyzed (Participants) | 161 | 145
  1 M, FU, no B-sy | 141 | 116
  1 M, FU, one B-sy: number analyzed (Participants) | 161 | 145
  1 M, FU, one B-sy | 20 | 29
  3 M, FU, no B-sy: number analyzed (Participants) | 153 | 119
  3 M, FU, no B-sy | 136 | 105
  3 M, FU, one B-sy: number analyzed (Participants) | 153 | 119
  3 M, FU, one B-sy | 17 | 14
  6 M, FU, no B-sy: number analyzed (Participants) | 138 | 107
  6 M, FU, no B-sy | 123 | 96
  6 M, FU, one B-sy: number analyzed (Participants) | 138 | 107
  6 M, FU, one B-sy | 15 | 11
  9 M, FU, no B-sy: number analyzed (Participants) | 129 | 96
  9 M, FU, no B-sy | 116 | 87
  9 M, FU, one B-sy: number analyzed (Participants) | 129 | 96
  9 M, FU, one B-sy | 13 | 9
  12 M, FU, no B-sy: number analyzed (Participants) | 119 | 87
  12 M, FU, no B-sy | 108 | 74
  12 M, FU, one B-sy: number analyzed (Participants) | 119 | 87
  12 M, FU, one B-sy | 11 | 13
  15 M, FU, no B-sy: number analyzed (Participants) | 103 | 71
  15 M, FU, no B-sy | 98 | 63
  15 M, FU, one B-sy: number analyzed (Participants) | 103 | 71
  15 M, FU, one B-sy | 5 | 8
  18 M, FU, no B-sy: number analyzed (Participants) | 98 | 64
  18 M, FU, no B-sy | 93 | 58
  18 M, FU, one B-sy: number analyzed (Participants) | 98 | 64
  18 M, FU, one B-sy | 5 | 6
  21 M, FU, no B-sy: number analyzed (Participants) | 94 | 60
  21 M, FU, no B-sy | 87 | 55
  21 M, FU, one B-sy: number analyzed (Participants) | 94 | 60
  21 M, FU, one B-sy | 7 | 5
  24 M, FU, no B-sy: number analyzed (Participants) | 80 | 52
  24 M, FU, no B-sy | 79 | 48
  24 M, FU, one B-sy: number analyzed (Participants) | 80 | 52
  24 M, FU, one B-sy | 1 | 4
  27 M, FU, no B-sy: number analyzed (Participants) | 74 | 45
  27 M, FU, no B-sy | 71 | 41
  27 M, FU, one B-syn: number analyzed (Participants) | 74 | 45
  27 M, FU, one B-syn | 4 | 3
  30 M, FU, no B-sy: number analyzed (Participants) | 70 | 35
  30 M, FU, no B-sy | 68 | 33
  30 M, FU, one B-sy: number analyzed (Participants) | 70 | 35
  30 M, FU, one B-sy | 2 | 2
  33 M, FU, no B-sy: number analyzed (Participants) | 66 | 29
  33 M, FU, no B-sy | 63 | 27
  33 M, FU, one B-sy: number analyzed (Participants) | 66 | 29
  33 M, FU, one B-sy | 3 | 2
  36 M, FU, no B-sy: number analyzed (Participants) | 58 | 23
  36 M, FU, no B-sy | 56 | 23
  36 M, FU, one B-sy: number analyzed (Participants) | 58 | 23
  36 M, FU, one B-sy | 2 | 0
  39 M, FU, no B-sy: number analyzed (Participants) | 52 | 18
  39 M, FU, no B-sy | 49 | 18
  39 M, FU, one B-sy: number analyzed (Participants) | 52 | 18
  39 M, FU, one B-sy | 3 | 0
  42 M, FU, no B-sy: number analyzed (Participants) | 45 | 16
  42 M, FU, no B-sy | 45 | 16
  42 M, FU, one B-sy: number analyzed (Participants) | 45 | 16
  42 M, FU, one B-sy | 0 | 0
  45 M, FU, no B-sy: number analyzed (Participants) | 41 | 15
  45 M, FU, no B-sy | 41 | 14
  45 M, FU, one B-sy: number analyzed (Participants) | 41 | 15
  45 M, FU, one B-sy | 0 | 1
  48 M, FU, no B-sy: number analyzed (Participants) | 37 | 13
  48 M, FU, no B-sy | 36 | 13
  48 M, FU, one B-sy: number analyzed (Participants) | 37 | 13
  48 M, FU, one B-sy | 1 | 0
  51 M, FU, no B-sy: number analyzed (Participants) | 32 | 12
  51 M, FU, no B-sy | 32 | 11
  51 M, FU, one B-sy: number analyzed (Participants) | 32 | 12
  51 M, FU, one B-sy | 0 | 1
  54 M, FU, no B-sy: number analyzed (Participants) | 30 | 10
  54 M, FU, no B-sy | 30 | 10
  54 M, FU, one B-sy: number analyzed (Participants) | 30 | 10
  54 M, FU, one B-sy | 0 | 0
  57 M, FU, no B-sy: number analyzed (Participants) | 26 | 9
  57 M, FU, no B-sy | 26 | 9
  57 M, FU, one B-sy: number analyzed (Participants) | 26 | 9
  57 M, FU, one B-sy | 0 | 0
  60 M, FU, no B-sy: number analyzed (Participants) | 25 | 9
  60 M, FU, no B-sy | 24 | 9
  60 M, FU, one B-sy: number analyzed (Participants) | 25 | 9
  60 M, FU, one B-sy | 1 | 0

9. Secondary Outcome: Percentage of Participants With the Best Overall Response (OR), as Assessed by the IRC
Description: OR is defined as the number of participants achieving an objective response (complete response [CR], CR with incomplete bone marrow recovery [CRi], partial response [PR], and nodular PR [nPR]). CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM.
Time Frame: From randomization up to 5 years after last dose of study drug
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Percentage of participants
  CR | 27 | 7
  CRi | 2 | 1
  nPR | 0 | 0
  PR | 55 | 59
  Stable disease | 11 | 28
  Progressive Disease | 0 | 0
  Not Evaluable | 4 | 2
  Missing | 1 | 2
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel

10. Secondary Outcome: Percentage of Participants With the Best OR, as Assessed by the Investigator
Description: OR is defined as the number of participants achieving an objective response (complete response [CR], CR with incomplete bone marrow recovery [CRi], partial response [PR], and nodular PR [nPR]). CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM.
  Responder = CR + CRi + NPR + PR
Time Frame: From randomization up to 5 years after last dose of study drug
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Percentage of participants
  CR | 45 | 24
  CRi | 12 | 4
  nPR | 2 | 8
  PR | 107 | 113
  Stable disease | 9 | 21
  Progressive Disease | 0 | 3
  Missing | 8 | 9
  Responder | 166 | 149
Statistical Analysis 1: Comparison: Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects vs Fludarabine + Cyclophosphamide_ ITT Subjects; Test type: Superiority or Other; p = 0.0166, Cochran-Mantel-Haenszel

11. Secondary Outcome: Number of Participants Who Were Negative for Minimal Residual Disease (MRD) Assessed by IRC
Description: MRD refers to small number of leukemic cells that remain in the participant during treatment or after treatment at the time the participant achieved a confirmed CR. MRD analysis was performed for the participants who were suspected of achieving a primary endpoint CR. MDR was performed by flow cytometry on a bone marrow or peripheral blood sample taken at least 2 months after final treatment. MRD negative was defined as less than one CLL cell per 10000 leukocytes.
Time Frame: From randomization up to 5 years after last dose of study drug
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Participants
  Screening: number analyzed (Participants) | 46 | 13
  Screening | 0 | 0
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 0
  Cycle 1 Day 1 | 0 |
  3 M, FU: number analyzed (Participants) | 44 | 12
  3 M, FU | 21 | 7
  6 M, FU: number analyzed (Participants) | 35 | 11
  6 M, FU | 25 | 6
  9 M, FU: number analyzed (Participants) | 29 | 8
  9 M, FU | 20 | 4
  12 M, FU: number analyzed (Participants) | 25 | 4
  12 M, FU | 16 | 1
  15 M, FU: number analyzed (Participants) | 20 | 3
  15 M, FU | 14 | 1
  18 M, FU: number analyzed (Participants) | 16 | 2
  18 M, FU | 12 | 1
  21 M, FU: number analyzed (Participants) | 13 | 2
  21 M, FU | 9 | 1
  24 M, FU: number analyzed (Participants) | 9 | 2
  24 M, FU | 8 | 1
  27 M, FU: number analyzed (Participants) | 9 | 1
  27 M, FU | 8 | 0
  30 M, FU: number analyzed (Participants) | 9 | 2
  30 M, FU | 8 | 2
  33 M, FU: number analyzed (Participants) | 5 | 2
  33 M, FU | 3 | 1
  36 M, FU: number analyzed (Participants) | 5 | 2
  36 M, FU | 5 | 1
  39 M, FU: number analyzed (Participants) | 2 | 1
  39 M, FU | 2 | 1
  42 M, FU: number analyzed (Participants) | 2 | 0
  42 M, FU | 2 |
  45 M, FU: number analyzed (Participants) | 1 | 1
  45 M, FU | 1 | 1
  48 M, FU: number analyzed (Participants) | 2 | 1
  48 M, FU | 2 | 1
  51 M, FU: number analyzed (Participants) | 2 | 1
  51 M, FU | 2 | 1
  54 M, FU: number analyzed (Participants) | 2 | 1
  54 M, FU | 2 | 1

12. Secondary Outcome: Number of Participants Who Were Negative for MRD Assessed by Investigator
Description: as for outcome 11
Time Frame: From randomization up to 5 years after last dose of study drug
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Participants
  Screening: number analyzed (Participants) | 177 | 171
  Screening | 0 | 1
  3 M, FU: number analyzed (Participants) | 120 | 76
  3 M, FU | 39 | 15
  6 M, FU: number analyzed (Participants) | 87 | 57
  6 M, FU | 48 | 11
  9 M, FU: number analyzed (Participants) | 71 | 29
  9 M, FU | 35 | 6
  12 M, FU: number analyzed (Participants) | 55 | 18
  12 M, FU | 31 | 3
  15 M, FU: number analyzed (Participants) | 38 | 14
  15 M, FU | 23 | 2
  18 M, FU: number analyzed (Participants) | 31 | 13
  18 M, FU | 20 | 2
  21 M, FU: number analyzed (Participants) | 27 | 9
  21 M, FU | 16 | 3
  24 M, FU: number analyzed (Participants) | 15 | 4
  24 M, FU | 13 | 2
  27 M, FU: number analyzed (Participants) | 18 | 5
  27 M, FU | 14 | 1
  30 M, FU: number analyzed (Participants) | 15 | 3
  30 M, FU | 12 | 3
  33 M, FU: number analyzed (Participants) | 13 | 3
  33 M, FU | 8 | 2
  36 M, FU: number analyzed (Participants) | 10 | 4
  36 M, FU | 9 | 2
  39 M, FU: number analyzed (Participants) | 7 | 3
  39 M, FU | 6 | 2
  42 M, FU: number analyzed (Participants) | 8 | 1
  42 M, FU | 7 | 1
  45 M, FU: number analyzed (Participants) | 7 | 2
  45 M, FU | 6 | 2
  48 M, FU: number analyzed (Participants) | 6 | 3
  48 M, FU | 6 | 2
  51 M, FU: number analyzed (Participants) | 6 | 2
  51 M, FU | 5 | 1
  54 M, FU: number analyzed (Participants) | 7 | 2
  54 M, FU | 4 | 2
  57 M, FU: number analyzed (Participants) | 4 | 3
  57 M, FU | 3 | 2
  60 M, FU: number analyzed (Participants) | 3 | 3
  60 M, FU | 3 | 2

13. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury.
Time Frame: From first dose of study medication to 60 Days after the last dose of study medication (for an AE), or up to 5 years after the last dose of study drug or until the time of the next anti-CLL therapy (for SAE)
Population: Safety Population: Participants who received at least one dose of a study drug.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Participants
  AE | 170 | 153
  SAE | 108 | 86

14. Secondary Outcome: Number of Participants With a Human Anti-human Antibody (HAHA) Positive Result at Indicated Time Points
Description: Serum samples for analysis of HAHA were collected at Baseline (Screening), after 3 cycles were compelted, after 1 M and 6 M post last dose. All samples were first tested in a screening step; positive samples from the screening were further evaluated in a confirmation test. The confirmed positive samples were reported as HAHA-positive.
Time Frame: From start of study drug until 60 days after the last dose of study medication
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles)
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Participants
  Screening Visit, n= 179,177: number analyzed (Participants) | 179 | 177
  Screening Visit, n= 179,177 | 8 | 1
  Cycle 4 Day 1, n= 151,130: number analyzed (Participants) | 151 | 130
  Cycle 4 Day 1, n= 151,130 | 0 | 2
  1 M, FU, n= 148,132: number analyzed (Participants) | 148 | 132
  1 M, FU, n= 148,132 | 0 | 2
  3 M, FU, n= 0,1: number analyzed (Participants) | 0 | 1
  3 M, FU, n= 0,1 |  | 0
  6 M, FU, n= 130, 99: number analyzed (Participants) | 130 | 99
  6 M, FU, n= 130, 99 | 2 | 0
  9 M, FU, n= 0, 2: number analyzed (Participants) | 0 | 2
  9 M, FU, n= 0, 2 |  | 0
  30 M, FU, n= 2, 0: number analyzed (Participants) | 2 | 0
  30 M, FU, n= 2, 0 | 0 |

15. Secondary Outcome: Number of Participants With Autoimmune Hemolytic Anaemia (AIHA)
Description: AIHA is a condition where the body's immune system fails to recognize red blood cells as "self" and begins destroying these red blood cells. The number of participants experienced AIHA are presented.
Time Frame: as for outcome 13
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Participants | 3 | 2

16. Secondary Outcome: Number of Participants With Drug Related Infections Reported as AEs and SAEs of Maximum Severity of Grade 3 or Higher
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Maximum severity grades were evaluated according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: as for outcome 13
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Participants
  AE | 19 | 11
  SAE | 25 | 21

17. Secondary Outcome: Number of Participants With at Least One Grade 3/Grade 4 Myelosuppression Adverse Events
Description: Participants with at least one Grade 3 or Grade 4 myelosuppression (anemia, neutropenia, and thrombocytopenia) are presented. Myelosuppression is defined as the decrease in the ability of the bone marrow to produce blood cells. AEs were graded according to NCI common terminology criteria for adverse events (CTCAE) grade, version 3.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: as for outcome 13
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Participants | 126 | 118

18. Secondary Outcome: Number of Participants Who Received no Transfusion or at Least One Transfusion During the Study
Description: Participants who received no transfusion and at least one transfusion during the study are presented. Participants who took any blood products or blood supportive care product are included.
Time Frame: From randomization up to 5 years after last dose of study drug
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Participants
  At least one transfusion | 125 | 99
  No transfusions | 56 | 79

19. Secondary Outcome: Mean Level of Immunoglobulin (Ig) Antibodies IgA, IgG, and IgM
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. Blood samples were collected from each participant and IgA, IgG, and IgM were measured at Baseline, and 1M and 6M after last dose during follow up period.
Time Frame: Baseline, 1M and 6M follow up
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
Gram per liter
  Cycle 1 Day 1, IgA: number analyzed (Participants) | 179 | 175
  Cycle 1 Day 1, IgA | 1.0 (0.74) | 0.9 (0.68)
  Cycle 1 Day 1, IgG: number analyzed (Participants) | 179 | 175
  Cycle 1 Day 1, IgG | 8.7 (5.22) | 8.2 (3.86)
  Cycle 1 Day 1, IgM: number analyzed (Participants) | 179 | 175
  Cycle 1 Day 1, IgM | 0.6 (1.36) | 0.8 (1.77)
  1 M, FU, IgA: number analyzed (Participants) | 150 | 131
  1 M, FU, IgA | 1.0 (0.79) | 1.0 (0.77)
  1 M, FU, IgG: number analyzed (Participants) | 150 | 131
  1 M, FU, IgG | 7.9 (4.05) | 7.9 (3.38)
  1 M, FU, IgM: number analyzed (Participants) | 150 | 131
  1 M, FU, IgM | 0.5 (1.16) | 0.8 (1.88)
  6 M, FU, IgA: number analyzed (Participants) | 130 | 101
  6 M, FU, IgA | 1.0 (0.77) | 1.0 (0.76)
  6 M, FU, IgG: number analyzed (Participants) | 130 | 101
  6 M, FU, IgG | 7.8 (3.97) | 8.9 (4.31)
  6 M, FU, IgM: number analyzed (Participants) | 130 | 101
  6 M, FU, IgM | 0.4 (0.50) | 1.1 (1.98)
  9 M, FU, IgA: number analyzed (Participants) | 1 | 2
  9 M, FU, IgA | 0.9 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. | 0.9 (0.21)
  9 M, FU, IgG: number analyzed (Participants) | 1 | 2
  9 M, FU, IgG | 15.2 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. | 8.8 (6.87)
  9 M, FU, IgM: number analyzed (Participants) | 1 | 2
  9 M, FU, IgM | 0.8 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. | 0.2 (0.04)
  18 M, FU, IgA: number analyzed (Participants) | 0 | 1
  18 M, FU, IgA |  | 2.4 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  18 M, FU, IgG: number analyzed (Participants) | 0 | 1
  18 M, FU, IgG |  | 9.1 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  18 M, FU, IgM: number analyzed (Participants) | 0 | 1
  18 M, FU, IgM |  | 1.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  30 M, FU, IgA: number analyzed (Participants) | 2 | 0
  30 M, FU, IgA | 1.3 (1.17) |
  30 M, FU, IgG: number analyzed (Participants) | 2 | 0
  30 M, FU, IgG | 4.7 (0.33) |
  30 M, FU, IgM: number analyzed (Participants) | 2 | 0
  30 M, FU, IgM | 0.4 (0.26) |

20. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) Cell Counts, CD5+ and CD19+
Description: CD5+ and CD19+ cells were counted by flow cytometry at Screening (Baseline) on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 during the treatment period and after last dose of study drug at 1 M and then every three month follow up up to 45 M. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus. Baseline is defined as the assessment closest to but prior to first dose (e.g. day 1 if available, otherwise, screening). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Screening, Cycle 1 Day1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 and after last dose at 1 M and then every three months up to 45 M during Follow-up Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
cells/uL
  Cycle 1 Day 1: number analyzed (Participants) | 71 | 65
  Cycle 1 Day 1 | 43180.6 (48784.64) | 53208.7 (70944.56)
  Cycle 1 Day 15: number analyzed (Participants) | 69 | 62
  Cycle 1 Day 15 | 2656.9 (6418.02) | 9244.0 (19610.62)
  Cycle 2 Day 1: number analyzed (Participants) | 68 | 63
  Cycle 2 Day 1 | 2057.4 (5525.72) | 10318.8 (21453.15)
  Cycle 2 Day 15: number analyzed (Participants) | 68 | 59
  Cycle 2 Day 15 | 513.7 (1717.65) | 6874.4 (20632.64)
  Cycle 3 Day 1: number analyzed (Participants) | 68 | 59
  Cycle 3 Day 1 | 790.0 (2953.42) | 6423.6 (19725.57)
  Cycle 4 Day 1: number analyzed (Participants) | 62 | 49
  Cycle 4 Day 1 | 402.1 (1768.74) | 2643.2 (8092.22)
  Cycle 5 Day 1: number analyzed (Participants) | 57 | 45
  Cycle 5 Day 1 | 142.6 (472.24) | 2838.6 (8314.08)
  Cycle 6 Day 1: number analyzed (Participants) | 56 | 39
  Cycle 6 Day 1 | 109.8 (398.77) | 3862.7 (13312.14)
  1 M, FU: number analyzed (Participants) | 64 | 61
  1 M, FU | 163.5 (685.41) | 5514.3 (17369.97)
  3 M, FU: number analyzed (Participants) | 69 | 47
  3 M, FU | 671.3 (2786.99) | 2604.9 (9229.90)
  6 M, FU: number analyzed (Participants) | 61 | 42
  6 M, FU | 1591.6 (8857.22) | 2275.6 (5118.00)
  9 M, FU: number analyzed (Participants) | 56 | 37
  9 M, FU | 910.5 (2495.85) | 3408.4 (7438.45)
  12 M, FU: number analyzed (Participants) | 47 | 30
  12 M, FU | 2303.2 (6675.70) | 2876.5 (6252.53)
  15 M, FU: number analyzed (Participants) | 35 | 18
  15 M, FU | 3325.8 (8006.48) | 3072.7 (9038.23)
  18 M, FU: number analyzed (Participants) | 22 | 12
  18 M, FU | 1607.5 (2935.82) | 4549.8 (8839.23)
  21 M, FU: number analyzed (Participants) | 22 | 10
  21 M, FU | 3830.8 (8989.02) | 5236.9 (10537.31)
  24 M, FU: number analyzed (Participants) | 9 | 6
  24 M, FU | 1244.6 (1300.01) | 7843.3 (11897.55)
  27 M, FU: number analyzed (Participants) | 7 | 4
  27 M, FU | 1877.4 (2117.84) | 6128.0 (9161.38)
  30 M, FU: number analyzed (Participants) | 6 | 2
  30 M, FU | 5029.7 (8266.90) | 6515.5 (5916.36)
  33 M, FU: number analyzed (Participants) | 4 | 1
  33 M, FU | 14166.8 (20166.09) | 5208.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  36 M, FU: number analyzed (Participants) | 3 | 1
  36 M, FU | 1187.0 (1407.79) | 8184.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  39 M, FU: number analyzed (Participants) | 1 | 0
  39 M, FU | 557.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. |
  42 M, FU: number analyzed (Participants) | 1 | 0
  42 M, FU | 1640.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. |
  45 M, FU: number analyzed (Participants) | 2 | 0
  45 M, FU | 4689.0 (1493.41) |
  48 M FU: number analyzed (Participants) | 1 | 1
  48 M FU | 27755.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. | 29155.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  54 M FU: number analyzed (Participants) | 1 | 0
  54 M FU | 189849.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. |

21. Secondary Outcome: Change From Baseline in Cell Counts, CD5- CD19+
Description: CD5- CD19+ cells were counted by flow cytometry at Screening (baseline) at Cycle 1 Day1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 during treatment period and after last dose of study drug at 1 M and then every three month up to 45 M during follow up period. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus. Baseline is defined as the assessment closest to but prior to first dose (e.g. Day 1 if available otherwise screening). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Screening, Cycle 1 Day1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 and after last dose at 1 M and then every three month up to 45 M during Follow-up Period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 181 | 178
cells/uL
  Screening: number analyzed (Participants) | 71 | 62
  Screening | 4817.8 (20948.17) | 6959.1 (39980.14)
  Cycle 1 Day 1: number analyzed (Participants) | 71 | 65
  Cycle 1 Day 1 | 5996.7 (22331.29) | 2041.3 (4418.63)
  Cycle 1 Day 15: number analyzed (Participants) | 69 | 62
  Cycle 1 Day 15 | 239.0 (1052.19) | 351.7 (1377.56)
  Cycle 2 Day 1: number analyzed (Participants) | 68 | 63
  Cycle 2 Day 1 | 115.4 (403.09) | 465.7 (1610.05)
  Cycle 2 Day 15: number analyzed (Participants) | 68 | 59
  Cycle 2 Day 15 | 35.6 (133.75) | 331.3 (1177.18)
  Cycle 3 Day 1: number analyzed (Participants) | 68 | 59
  Cycle 3 Day 1 | 39.5 (144.64) | 179.7 (520.63)
  Cycle 4 Day 1: number analyzed (Participants) | 62 | 49
  Cycle 4 Day 1 | 25.7 (92.88) | 95.3 (369.19)
  Cycle 5 Day 1: number analyzed (Participants) | 57 | 45
  Cycle 5 Day 1 | 15.9 (77.11) | 195.5 (945.34)
  Cycle 6 Day 1: number analyzed (Participants) | 56 | 39
  Cycle 6 Day 1 | 10.0 (29.85) | 649.7 (3606.28)
  1 M, FU: number analyzed (Participants) | 64 | 61
  1 M, FU | 7.5 (19.54) | 863.8 (5001.84)
  3 M, FU: number analyzed (Participants) | 69 | 47
  3 M, FU | 40.1 (238.18) | 172.0 (681.28)
  6 M, FU: number analyzed (Participants) | 61 | 42
  6 M, FU | 21.2 (58.16) | 50.7 (49.13)
  9 M, FU: number analyzed (Participants) | 56 | 37
  9 M, FU | 85.7 (359.01) | 92.0 (101.16)
  12 M, FU: number analyzed (Participants) | 47 | 30
  12 M, FU | 89.9 (226.06) | 220.1 (698.57)
  15 M, FU: number analyzed (Participants) | 35 | 18
  15 M, FU | 67.3 (59.52) | 94.6 (70.17)
  18 M, FU: number analyzed (Participants) | 22 | 12
  18 M, FU | 126.1 (188.25) | 92.3 (69.14)
  21 M, FU: number analyzed (Participants) | 22 | 10
  21 M, FU | 375.5 (1307.35) | 108.3 (95.86)
  24 M, FU: number analyzed (Participants) | 9 | 6
  24 M, FU | 74.0 (57.46) | 104.5 (70.46)
  27 M, FU: number analyzed (Participants) | 7 | 4
  27 M, FU | 73.9 (60.40) | 187.5 (200.85)
  30 M, FU: number analyzed (Participants) | 6 | 2
  30 M, FU | 74.2 (58.82) | 129.5 (5303)
  33 M, FU: number analyzed (Participants) | 4 | 1
  33 M, FU | 41.8 (40.13) | 1003.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  36 M, FU: number analyzed (Participants) | 3 | 1
  36 M, FU | 107.3 (86.75) | 1506.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  39 M, FU: number analyzed (Participants) | 1 | 0
  39 M, FU | 13.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. |
  42 M, FU: number analyzed (Participants) | 1 | 0
  42 M, FU | 13.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. |
  45 M, FU: number analyzed (Participants) | 2 | 0
  45 M, FU | 166.5 (222.74) |
  48 M, FU: number analyzed (Participants) | 1 | 1
  48 M, FU | 6528.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. | 28.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed.
  54 M, FU: number analyzed (Participants) | 1 | 0
  54 M, FU | 690.0 (NA) — No standard deviation was able to be calculated for this data point because only one participant was analyzed. |

22. Secondary Outcome: Prognostic and Biological Markers Correlating With Clinical Response
Description: Blood samples were collected for the assessment of the following prognostic markers at BL: immunoglobulin heavy chain variable region(IgVH) homology; Zeta-Chain-Associated Protein Kinase 70(ZAP70), VH3-21 usage; Cytogenetics (by fluorescent in situ hybridization [FISH]); beta 2 microglobulin. Cox-regression model was used to explore the relationship between progression-free survival and the following explanatory variables: treatment group, cytogenetics (analyzed by FISH included 6q-,11q-, +12q, 17p-, 13q-) , ZAP-70 (positive, negative or intermediate), VH3-21 usage (Yes and No), IgVH homology (>98%, 97%-98% and <97%), beta 2 microglobulin (>3500 microgram per liter [µg/L] and <=3500 µg/L). For each covariate, a hazard ratio <1 indicates a lower risk on the first effect tested compared with the other effects tested. Cytogenetics Group (based on >=20%)=cytogenetics (CY G).
Time Frame: From randomization up to 5 years after last dose of study drug
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Participants
  B2 Microglobulin G 1: > 3500 microgram/liter (μg/L | 79 | 78
  B2 Microglobulin G 1: <= 3500 ug/L: number analyzed (Participants) | 51 | 47
  B2 Microglobulin G 1: <= 3500 ug/L | 22 | 26
  CY G 1: 11q-: number analyzed (Participants) | 40 | 31
  CY G 1: 11q- | 29 | 19
  CY G 1: 17p-: number analyzed (Participants) | 7 | 13
  CY G 1: 17p- | 6 | 9
  CY G 1: 6q- or +12q or 13q-: number analyzed (Participants) | 84 | 80
  CY G 1: 6q- or +12q or 13q- | 38 | 48
  CY G 1: no aberration: number analyzed (Participants) | 45 | 47
  CY G 1: no aberration | 27 | 27
  VH3-21 Usage Flag: Yes: number analyzed (Participants) | 9 | 7
  VH3-21 Usage Flag: Yes | 6 | 4
  VH3-21 Usage Flag: No: number analyzed (Participants) | 159 | 162
  VH3-21 Usage Flag: No | 93 | 96
  IgVH Homology, <97%: number analyzed (Participants) | 40 | 43
  IgVH Homology, <97% | 13 | 15
  IgVH Homology, 97%-98%: number analyzed (Participants) | 12 | 10
  IgVH Homology, 97%-98% | 5 | 7
  IgVH Homology, >98%: number analyzed (Participants) | 115 | 116
  IgVH Homology, >98% | 80 | 78
  ZAP70 G 1, Negative: number analyzed (Participants) | 28 | 32
  ZAP70 G 1, Negative | 14 | 13
  ZAP70 G 1, Intermediate: number analyzed (Participants) | 54 | 46
  ZAP70 G 1, Intermediate | 27 | 23
  ZAP70, G1 Positive: number analyzed (Participants) | 94 | 91
  ZAP70, G1 Positive | 60 | 65

23. Secondary Outcome: Changes in Patient Reported Outcome (PRO) Measures and Scores for European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Chronic Lymphocytic Leukaemia 16 Item Module (EORTC QLQ-CLL 16)
Description: The EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life (HRQoL) important in CLL. There are 4 multi-item scales - fatigue (2 items), treatment side effects ([TSE], 4 items), disease symptoms (disease effects scale [DES], 4 items), and infection scale [IS] (4 items) - and single item scales (social activities [Social Problems (SP) Scale] and future health worries[Future Health (FH) Scale].). These are measured on a four point scale where 1 = not at all and 4 = very much. These scores are transformed to give a rating from 0 - 100, where 0 =no symptoms or problems and 100 = a severe symptoms or problems. EORTC QLQ-CLL16 was assessed at Screening; Cycle 4 Day 1 and during follow-up 1 M and every 3 M up to 24 months. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value was obtained at randomization.
Time Frame: Screening, Cycle 3 Day 1, and 1 M and every 3 month post last dose up to 24 month.
Population: Participants
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
scores on a scale
  DES, Cycle 4 Day 1: number analyzed (Participants) | 142 | 125
  DES, Cycle 4 Day 1 | -8.5 (18.08) | -9.0 (17.16)
  DES, 1 M, FU: number analyzed (Participants) | 138 | 123
  DES, 1 M, FU | -9.7 (19.18) | -9.8 (19.89)
  DES, 3 M, FU: number analyzed (Participants) | 145 | 109
  DES, 3 M, FU | -8.2 (19.48) | -10.9 (19.07)
  DES, 6 M, FU: number analyzed (Participants) | 126 | 99
  DES, 6 M, FU | -9.8 (17.99) | -11.6 (18.05)
  DES, 9 M, FU: number analyzed (Participants) | 115 | 85
  DES, 9 M, FU | -8.2 (20.70) | -12.0 (17.04)
  DES. 12 M, FU: number analyzed (Participants) | 109 | 76
  DES. 12 M, FU | -10.1 (18.64) | -10.2 (16.09)
  DES, 15 M, FU: number analyzed (Participants) | 98 | 62
  DES, 15 M, FU | -8.6 (18.08) | -10.2 (16.91)
  DES, 18 M, FU: number analyzed (Participants) | 90 | 59
  DES, 18 M, FU | -8.5 (18.53) | -11.6 (18.79)
  DES, 21 M, FU: number analyzed (Participants) | 87 | 53
  DES, 21 M, FU | -8.2 (18.48) | -11.3 (17.60)
  DES, 24 M, FU: number analyzed (Participants) | 70 | 50
  DES, 24 M, FU | -7.1 (19.93) | -13.6 (16.18)
  Fatigue Scale (FS), Cycle 4 Day 1: number analyzed (Participants) | 142 | 125
  Fatigue Scale (FS), Cycle 4 Day 1 | -7.0 (22.57) | -7.1 (24.16)
  FS, 1 M, FU: number analyzed (Participants) | 139 | 123
  FS, 1 M, FU | -5.4 (29.16) | -6.2 (28.74)
  FS, 3 M, FU: number analyzed (Participants) | 144 | 109
  FS, 3 M, FU | -4.4 (26.30) | -8.3 (30.14)
  FS, 6 M, FU: number analyzed (Participants) | 126 | 99
  FS, 6 M, FU | -7.1 (25.94) | -12.0 (25.98)
  FS, 9 M, FU: number analyzed (Participants) | 115 | 85
  FS, 9 M, FU | -6.2 (27.08) | -10.6 (26.95)
  FS. 12 M, FU: number analyzed (Participants) | 109 | 76
  FS. 12 M, FU | -7.3 (27.26) | -8.1 (25.75)
  FS, 15 M, FU: number analyzed (Participants) | 97 | 62
  FS, 15 M, FU | -7.6 (22.57) | -9.9 (24.04)
  FS, 18 M, FU: number analyzed (Participants) | 90 | 59
  FS, 18 M, FU | -7.0 (23.03) | -3.7 (33.34)
  FS, 21 M, FU: number analyzed (Participants) | 87 | 53
  FS, 21 M, FU | -10.3 (24.28) | -8.2 (27.27)
  FS, 24 M, FU: number analyzed (Participants) | 69 | 50
  FS, 24 M, FU | -8.7 (24.19) | -8.7 (25.48)
  FH, Cycle 4 Day 1: number analyzed (Participants) | 141 | 123
  FH, Cycle 4 Day 1 | -11.8 (32.89) | -10.6 (27.76)
  FH, 1 M, FU: number analyzed (Participants) | 139 | 120
  FH, 1 M, FU | -15.3 (35.04) | -11.9 (29.56)
  FH, 3 M, FU: number analyzed (Participants) | 145 | 107
  FH, 3 M, FU | -14.3 (33.96) | -14.0 (32.06)
  FH, 6 M, FU: number analyzed (Participants) | 126 | 96
  FH, 6 M, FU | -13.4 (33.98) | -17.7 (30.57)
  FH, 9 M, FU: number analyzed (Participants) | 113 | 81
  FH, 9 M, FU | -15.6 (33.65) | -13.2 (34.43)
  FH. 12 M, FU: number analyzed (Participants) | 109 | 74
  FH. 12 M, FU | -14.1 (32.80) | -14.9 (33.63)
  FH, 15 M, FU: number analyzed (Participants) | 98 | 61
  FH, 15 M, FU | -14.6 (29.14) | -14.2 (34.13)
  FH, 18 M, FU: number analyzed (Participants) | 90 | 58
  FH, 18 M, FU | -15.9 (31.69) | -18.4 (33.72)
  FH, 21 M, FU: number analyzed (Participants) | 87 | 52
  FH, 21 M, FU | -16.9 (28.70) | -15.4 (29.12)
  FH, 24 M, FU: number analyzed (Participants) | 70 | 49
  FH, 24 M, FU | -21.0 (29.58) | -17.7 (30.51)
  IS, Cycle 4 Day 1: number analyzed (Participants) | 142 | 125
  IS, Cycle 4 Day 1 | 0.5 (17.65) | -1.4 (18.23)
  IS, 1 M, FU: number analyzed (Participants) | 138 | 122
  IS, 1 M, FU | 2.9 (22.79) | 2.7 (24.06)
  IS, 3 M, FU: number analyzed (Participants) | 144 | 109
  IS, 3 M, FU | 0.8 (19.42) | 0.8 (20.99)
  IS, 6 M, FU: number analyzed (Participants) | 126 | 99
  IS, 6 M, FU | -1.2 (18.46) | -0.9 (20.40)
  IS, 9 M, FU: number analyzed (Participants) | 115 | 85
  IS, 9 M, FU | -1.4 (18.81) | 1.4 (22.45)
  IS. 12 M, FU: number analyzed (Participants) | 109 | 76
  IS. 12 M, FU | 0.4 (19.22) | 2.1 (20.92)
  IS, 15 M, FU: number analyzed (Participants) | 97 | 60
  IS, 15 M, FU | 0.5 (17.56) | 0.3 (18.79)
  IS, 18 M, FU: number analyzed (Participants) | 89 | 59
  IS, 18 M, FU | -2.0 (16.04) | 0.9 (19.04)
  IS, 21 M, FU: number analyzed (Participants) | 87 | 53
  IS, 21 M, FU | -2.5 (18.13) | 2.5 (22.09)
  IS, 24 M, FU: number analyzed (Participants) | 69 | 49
  IS, 24 M, FU | -0.5 (18.85) | 0.5 (21.34)
  SP Scale Cycle 4 Day 1: number analyzed (Participants) | 141 | 125
  SP Scale Cycle 4 Day 1 | 1.9 (25.44) | 0.3 (26.94)
  SP Scale, 1 M, FU: number analyzed (Participants) | 137 | 121
  SP Scale, 1 M, FU | 3.2 (34.51) | 0.0 (35.22)
  SP Scale, 3 M, FU: number analyzed (Participants) | 143 | 109
  SP Scale, 3 M, FU | -1.9 (33.04) | -4.3 (35.75)
  SP Scale, 6 M, FU: number analyzed (Participants) | 124 | 98
  SP Scale, 6 M, FU | -5.6 (31.73) | -10.9 (30.56)
  SP Scale, 9 M, FU: number analyzed (Participants) | 114 | 85
  SP Scale, 9 M, FU | -5.0 (30.15) | -11.0 (31.45)
  SP Scale. 12 M, FU: number analyzed (Participants) | 107 | 75
  SP Scale. 12 M, FU | -7.2 (31.06) | -7.6 (34.47)
  SP Scale, 15 M, FU: number analyzed (Participants) | 95 | 61
  SP Scale, 15 M, FU | -6.7 (30.21) | -13.7 (30.05)
  SP Scale, 18 M, FU: number analyzed (Participants) | 89 | 59
  SP Scale, 18 M, FU | -7.1 (31.57) | -8.5 (40.40)
  SP Scale, 21 M, FU: number analyzed (Participants) | 86 | 53
  SP Scale, 21 M, FU | -8.1 (31.07) | -7.5 (37.92)
  SP Scale, 24 M, FU: number analyzed (Participants) | 68 | 50
  SP Scale, 24 M, FU | -11.8 (24.27) | -8.7 (36.15)
  TSE, Cycle 4 Day 1: number analyzed (Participants) | 142 | 125
  TSE, Cycle 4 Day 1 | -4.7 (16.15) | -4.0 (16.78)
  TSE, 1 M, FU: number analyzed (Participants) | 139 | 123
  TSE, 1 M, FU | -5.0 (18.09) | -3.2 (19.08)
  TSE, 3 M, FU: number analyzed (Participants) | 145 | 109
  TSE, 3 M, FU | -3.7 (19.41) | -4.3 (17.03)
  TSE, 6 M, FU: number analyzed (Participants) | 126 | 99
  TSE, 6 M, FU | -6.0 (15.25) | -4.8 (16.96)
  TSE, 9 M, FU: number analyzed (Participants) | 115 | 85
  TSE, 9 M, FU | -4.3 (17.22) | -5.1 (16.38)
  TSE. 12 M, FU: number analyzed (Participants) | 109 | 76
  TSE. 12 M, FU | -5.2 (16.44) | -3.2 (13.94)
  TSE, 15 M, FU: number analyzed (Participants) | 98 | 62
  TSE, 15 M, FU | -4.0 (14.92) | -4.2 (13.73)
  TSE, 18 M, FU: number analyzed (Participants) | 90 | 60
  TSE, 18 M, FU | -4.4 (17.10) | -3.6 (19.18)
  TSE, 21 M, FU: number analyzed (Participants) | 87 | 54
  TSE, 21 M, FU | -4.7 (16.63) | -4.0 (15.91)
  TSE, 24 M, FU: number analyzed (Participants) | 70 | 50
  TSE, 24 M, FU | -5.4 (17.52) | -6.5 (14.12)

24. Secondary Outcome: Change From Baseline in Patient Reported Outcome (PRO) as Assessed by EuroQoL Five-Dimension (EQ-5D) Score at Indicated Visit
Description: EQ-5D is comprised of a 5-item health status measure and a visual analogue scale (VAS) and is used to generate two scores: the utility score and the thermometer score. The utility score measures mobility, self-care, usual activities, pain, discomfort, and anxiety/depression. Responses to each of the 5 health states are measured on a 3-point scale (level 1 = no problem; level 2 = some or moderate problem(s) and level 3 = unable, or extreme problems). Responses are typically converted into health utilities or valuations on a scale ranging from 0 (death) to 1 (perfect health). The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. A Negative health status describes health state worse than death.Baseline is the most recent, non-missing value prior to or on the first study drug dose date.
Time Frame: Screening, Cycle 3 Day 1, and 1 M and every 3 month post last dose up to 24 month.
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Score on a scale
  UT, Cycle 4 Day 1: number analyzed (Participants) | 136 | 121
  UT, Cycle 4 Day 1 | 0.0 (0.27) | 0.0 (0.21)
  UT, 1 M, FU: number analyzed (Participants) | 133 | 117
  UT, 1 M, FU | 0.1 (0.22) | 0.0 (0.28)
  UT, 3 M, FU: number analyzed (Participants) | 141 | 102
  UT, 3 M, FU | 0.0 (0.27) | 0.1 (0.23)
  UT, 6 M, FU: number analyzed (Participants) | 122 | 96
  UT, 6 M, FU | 0.1 (0.24) | 0.1 (0.24)
  UT, 9 M, FU: number analyzed (Participants) | 110 | 81
  UT, 9 M, FU | 0.1 (0.26) | 0.1 (0.24)
  UT. 12 M, FU: number analyzed (Participants) | 107 | 71
  UT. 12 M, FU | 0.1 (0.21) | 0.1 (0.22)
  UT, 15 M, FU: number analyzed (Participants) | 96 | 58
  UT, 15 M, FU | 0.0 (0.23) | 0.1 (0.24)
  UT, 18 M, FU: number analyzed (Participants) | 88 | 57
  UT, 18 M, FU | 0.1 (0.21) | 0.0 (0.34)
  UT, 21 M, FU: number analyzed (Participants) | 87 | 52
  UT, 21 M, FU | 0.1 (0.21) | 0.1 (0.26)
  UT, 24 M, FU: number analyzed (Participants) | 68 | 47
  UT, 24 M, FU | 0.1 (0.19) | 0.1 (0.28)
  VAS Cycle 4 Day 1: number analyzed (Participants) | 137 | 122
  VAS Cycle 4 Day 1 | 6.1 (17.68) | 5.6 (17.64)
  VAS, 1 M, FU: number analyzed (Participants) | 138 | 122
  VAS, 1 M, FU | 5.6 (20.73) | 5.9 (22.83)
  VAS, 3 M, FU: number analyzed (Participants) | 141 | 107
  VAS, 3 M, FU | 5.7 (19.92) | 9.6 (20.88)
  VAS, 6 M, FU: number analyzed (Participants) | 124 | 99
  VAS, 6 M, FU | 8.2 (18.84) | 11.1 (19.08)
  VAS, 9 M, FU: number analyzed (Participants) | 114 | 85
  VAS, 9 M, FU | 8.1 (18.33) | 11.9 (20.59)
  VAS. 12 M, FU: number analyzed (Participants) | 108 | 75
  VAS. 12 M, FU | 7.0 (21.93) | 10.3 (21.21)
  VAS, 15 M, FU: number analyzed (Participants) | 95 | 62
  VAS, 15 M, FU | 8.0 (17.52) | 13.1 (21.06)
  VAS, 18 M, FU: number analyzed (Participants) | 89 | 60
  VAS, 18 M, FU | 9.4 (17.86) | 11.1 (25.40)
  VAS, 21 M, FU: number analyzed (Participants) | 87 | 53
  VAS, 21 M, FU | 8.1 (16.42) | 11.3 (24.16)
  VAS, 24 M, FU: number analyzed (Participants) | 69 | 50
  VAS, 24 M, FU | 8.8 (19.50) | 15.2 (21.88)

25. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30, a self-reported, cancer-specific instrument assessing 15 domains: physical, role, emotional, cognitive and social functioning, pain,fatigue, nausea and vomiting, insomnia, loss of appetite, constipation, diarrhea, and dyspnea, financial difficulties and a global health status/quality of life (QOF). Functional and symptoms scales were measured on four point Likert scale where 1 = not at all and 4 = very much. Pat. assessed at Screening; Cycle 4 Day 1 and during follow-up 1 M and every 3 M up to 24 months. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Clinically meaningful changes or minimally important differences (MIDs)have been previously established for the EORTC QLQ C30, and categorized as 'small' if the mean change in scores is 5-10 points, 'moderate' if 10-20 points, and 'large' if >20points.
Time Frame: Screening, Cycle 3 Day 1, and 1 M and every 3 month post last dose up to 24 month.
Population: ITT Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Scores on a scale
  Appetite Loss, Cycle 4 Day 1: number analyzed (Participants) | 140 | 124
  Appetite Loss, Cycle 4 Day 1 | 0.5 (25.60) | -1.9 (26.65)
  Appetite Loss, 1 M, FU: number analyzed (Participants) | 136 | 119
  Appetite Loss, 1 M, FU | -0.2 (26.14) | -3.9 (28.52)
  Appetite Loss, 3 M, FU: number analyzed (Participants) | 142 | 108
  Appetite Loss, 3 M, FU | -0.7 (26.77) | -7.4 (28.22)
  Appetite Loss, 6 M, FU: number analyzed (Participants) | 123 | 97
  Appetite Loss, 6 M, FU | -6.0 (23.00) | -12.4 (26.05)
  Appetite Loss, 9 M, FU: number analyzed (Participants) | 112 | 83
  Appetite Loss, 9 M, FU | -3.9 (20.38) | -9.6 (25.25)
  Appetite Loss. 12 M, FU: number analyzed (Participants) | 107 | 72
  Appetite Loss. 12 M, FU | -4.0 (22.76) | -6.0 (27.59)
  Appetite Loss, 15 M, FU: number analyzed (Participants) | 96 | 60
  Appetite Loss, 15 M, FU | -3.8 (23.13) | -9.4 (28.19)
  Appetite Loss, 18 M, FU: number analyzed (Participants) | 89 | 60
  Appetite Loss, 18 M, FU | -7.9 (20.11) | -9.4 (30.12)
  Appetite Loss, 21 M, FU: number analyzed (Participants) | 87 | 52
  Appetite Loss, 21 M, FU | -3.4 (20.36) | -7.7 (27.70)
  Appetite Loss, 24 M, FU: number analyzed (Participants) | 69 | 48
  Appetite Loss, 24 M, FU | -3.9 (22.53) | -12.5 (29.68)
  Cognitive Functioning, Cycle 4 Day 1: number analyzed (Participants) | 142 | 126
  Cognitive Functioning, Cycle 4 Day 1 | 3.4 (18.25) | 2.5 (18.39)
  Cognitive Functioning, 1 M, FU: number analyzed (Participants) | 139 | 122
  Cognitive Functioning, 1 M, FU | -0.4 (18.40) | 3.0 (19.87)
  Cognitive Functioning, 3 M, FU: number analyzed (Participants) | 145 | 109
  Cognitive Functioning, 3 M, FU | 0.0 (18.74) | 2.3 (21.69)
  Cognitive Functioning, 6 M, FU: number analyzed (Participants) | 126 | 99
  Cognitive Functioning, 6 M, FU | 1.7 (18.95) | 2.7 (20.99)
  Cognitive Functioning, 9 M, FU: number analyzed (Participants) | 115 | 85
  Cognitive Functioning, 9 M, FU | -0.6 (20.58) | 2.4 (19.61)
  Cognitive Functioning. 12 M, FU: number analyzed (Participants) | 110 | 76
  Cognitive Functioning. 12 M, FU | -2.1 (19.17) | -1.8 (21.36)
  Cognitive Functioning, 15 M, FU: number analyzed (Participants) | 97 | 62
  Cognitive Functioning, 15 M, FU | -1.0 (17.97) | 0.3 (20.58)
  Cognitive Functioning, 18 M, FU: number analyzed (Participants) | 89 | 61
  Cognitive Functioning, 18 M, FU | -0.9 (20.00) | -0.3 (22.67)
  Cognitive Functioning, 21 M, FU: number analyzed (Participants) | 88 | 53
  Cognitive Functioning, 21 M, FU | -1.9 (21.65) | -1.9 (21.84)
  Cognitive Functioning, 24 M, FU: number analyzed (Participants) | 70 | 50
  Cognitive Functioning, 24 M, FU | 1.0 (20.83) | -1.3 (21.25)
  Constipation, Cycle 4 Day 1: number analyzed (Participants) | 142 | 126
  Constipation, Cycle 4 Day 1 | 2.1 (21.46) | 0.8 (18.60)
  Constipation, 1 M, FU: number analyzed (Participants) | 139 | 122
  Constipation, 1 M, FU | -0.7 (19.02) | 0.3 (18.92)
  Constipation, 3 M, FU: number analyzed (Participants) | 145 | 109
  Constipation, 3 M, FU | -2.1 (19.33) | -0.9 (20.01)
  Constipation, 6 M, FU: number analyzed (Participants) | 125 | 98
  Constipation, 6 M, FU | -3.5 (19.32) | 0.3 (18.22)
  Constipation, 9 M, FU: number analyzed (Participants) | 115 | 85
  Constipation, 9 M, FU | -1.2 (19.71) | 0.4 (18.18)
  Constipation. 12 M, FU: number analyzed (Participants) | 109 | 76
  Constipation. 12 M, FU | -0.0 (23.13) | 0.4 (19.24)
  Constipation, 15 M, FU: number analyzed (Participants) | 96 | 62
  Constipation, 15 M, FU | -1.7 (21.29) | -3.8 (20.11)
  Constipation, 18 M, FU: number analyzed (Participants) | 90 | 61
  Constipation, 18 M, FU | -0.4 (21.49) | -1.1 (24.32)
  Constipation, 21 M, FU: number analyzed (Participants) | 87 | 53
  Constipation, 21 M, FU | -1.9 (22.93) | -3.8 (23.26)
  Constipation, 24 M, FU: number analyzed (Participants) | 70 | 50
  Constipation, 24 M, FU | 0.0 (21.23) | -3.3 (21.56)
  Diarrhoea, Cycle 4 Day 1: number analyzed (Participants) | 141 | 125
  Diarrhoea, Cycle 4 Day 1 | 0.2 (19.72) | -2.4 (17.54)
  Diarrhoea, 1 M, FU: number analyzed (Participants) | 135 | 121
  Diarrhoea, 1 M, FU | -3.5 (20.87) | 0.8 (21.28)
  Diarrhoea, 3 M, FU: number analyzed (Participants) | 143 | 109
  Diarrhoea, 3 M, FU | 1.6 (22.49) | 1.5 (20.98)
  Diarrhoea, 6 M, FU: number analyzed (Participants) | 124 | 98
  Diarrhoea, 6 M, FU | 0.0 (20.38) | -3.1 (16.64)
  Diarrhoea, 9 M, FU: number analyzed (Participants) | 114 | 85
  Diarrhoea, 9 M, FU | 0.3 (20.56) | -2.7 (17.97)
  Diarrhoea. 12 M, FU: number analyzed (Participants) | 108 | 76
  Diarrhoea. 12 M, FU | -3.4 (15.75) | -2.2 (19.12)
  Diarrhoea, 15 M, FU: number analyzed (Participants) | 96 | 61
  Diarrhoea, 15 M, FU | -1.7 (19.57) | -4.4 (20.62)
  Diarrhoea, 18 M, FU: number analyzed (Participants) | 89 | 61
  Diarrhoea, 18 M, FU | -1.9 (17.67) | -1.1 (17.18)
  Diarrhoea, 21 M, FU: number analyzed (Participants) | 87 | 53
  Diarrhoea, 21 M, FU | -2.3 (18.88) | 0.6 (21.17)
  Diarrhoea, 24 M, FU: number analyzed (Participants) | 68 | 50
  Diarrhoea, 24 M, FU | -2.9 (17.02) | -0.7 (20.75)
  Dyspnoea Cycle 4 Day 1: number analyzed (Participants) | 138 | 124
  Dyspnoea Cycle 4 Day 1 | -4.6 (22.85) | -4.6 (23.41)
  Dyspnoea, 1 M, FU: number analyzed (Participants) | 139 | 121
  Dyspnoea, 1 M, FU | -1.0 (26.60) | -2.8 (25.67)
  Dyspnoea, 3 M, FU: number analyzed (Participants) | 141 | 108
  Dyspnoea, 3 M, FU | -3.1 (26.40) | -1.5 (25.53)
  Dyspnoea, 6 M, FU: number analyzed (Participants) | 124 | 97
  Dyspnoea, 6 M, FU | -2.7 (21.92) | -7.2 (24.17)
  Dyspnoea, 9 M, FU: number analyzed (Participants) | 113 | 83
  Dyspnoea, 9 M, FU | -2.7 (26.03) | -6.4 (23.55)
  Dyspnoea. 12 M, FU: number analyzed (Participants) | 108 | 73
  Dyspnoea. 12 M, FU | -3.4 (24.52) | -4.1 (22.87)
  Dyspnoea, 15 M, FU: number analyzed (Participants) | 95 | 60
  Dyspnoea, 15 M, FU | -2.5 (20.77) | -2.2 (26.66)
  Dyspnoea, 18 M, FU: number analyzed (Participants) | 90 | 59
  Dyspnoea, 18 M, FU | -3.0 (24.81) | -2.8 (29.22)
  Dyspnoea, 21 M, FU: number analyzed (Participants) | 87 | 52
  Dyspnoea, 21 M, FU | -3.4 (24.92) | -1.9 (21.30)
  Dyspnoea, 24 M, FU: number analyzed (Participants) | 69 | 49
  Dyspnoea, 24 M, FU | -2.4 (26.39) | -4.8 (24.53)
  Emotional Functioning Cycle 4 Day 1: number analyzed (Participants) | 142 | 125
  Emotional Functioning Cycle 4 Day 1 | 4.4 (17.91) | 5.4 (19.59)
  Emotional Functioning, 1 M, FU: number analyzed (Participants) | 139 | 122
  Emotional Functioning, 1 M, FU | 5.4 (20.26) | 7.2 (24.08)
  Emotional Functioning, 3 M, FU: number analyzed (Participants) | 145 | 109
  Emotional Functioning, 3 M, FU | 5.7 (20.93) | 7.8 (20.90)
  Emotional Functioning, 6 M, FU: number analyzed (Participants) | 126 | 99
  Emotional Functioning, 6 M, FU | 4.8 (22.57) | 8.9 (22.34)
  Emotional Functioning, 9 M: number analyzed (Participants) | 115 | 85
  Emotional Functioning, 9 M | 3.4 (22.95) | 6.7 (18.52)
  Emotional Functioning. 12 M, FU: number analyzed (Participants) | 110 | 76
  Emotional Functioning. 12 M, FU | 3.9 (22.11) | 8.0 (21.92)
  Emotional Functioning, 15 M, FU: number analyzed (Participants) | 98 | 62
  Emotional Functioning, 15 M, FU | 5.1 (21.54) | 6.5 (21.15)
  Emotional Functioning, 18 M, FU: number analyzed (Participants) | 90 | 61
  Emotional Functioning, 18 M, FU | 5.1 (22.94) | 6.5 (26.35)
  Emotional Functioning, 21 M, FU: number analyzed (Participants) | 88 | 52
  Emotional Functioning, 21 M, FU | 5.3 (22.43) | 7.7 (23.56)
  Emotional Functioning, 24 M, FU: number analyzed (Participants) | 70 | 50
  Emotional Functioning, 24 M, FU | 7.1 (23.02) | 7.1 (26.16)
  Fatigue Cycle 4 Day 1: number analyzed (Participants) | 142 | 126
  Fatigue Cycle 4 Day 1 | -4.3 (21.37) | -6.3 (22.66)
  Fatigue, 1 M, FU: number analyzed (Participants) | 138 | 122
  Fatigue, 1 M, FU | -7.4 (25.16) | -4.5 (28.64)
  Fatigue, 3 M, FU: number analyzed (Participants) | 145 | 109
  Fatigue, 3 M, FU | -5.4 (24.01) | -9.3 (27.83)
  Fatigue, 6 M, FU: number analyzed (Participants) | 126 | 99
  Fatigue, 6 M, FU | -8.2 (23.64) | -12.2 (22.43)
  Fatigue, 9 M, FU: number analyzed (Participants) | 115 | 86
  Fatigue, 9 M, FU | -8.8 (23.80) | -9.8 (24.56)
  Fatigue. 12 M, FU: number analyzed (Participants) | 110 | 76
  Fatigue. 12 M, FU | -6.8 (25.28) | -10.3 (23.44)
  Fatigue, 15 M, FU: number analyzed (Participants) | 97 | 76
  Fatigue, 15 M, FU | -7.6 (19.83) | -8.9 (27.61)
  Fatigue, 18 M, FU: number analyzed (Participants) | 90 | 62
  Fatigue, 18 M, FU | -7.0 (22.25) | -6.1 (30.15)
  Fatigue, 21 M, FU: number analyzed (Participants) | 88 | 53
  Fatigue, 21 M, FU | -9.6 (20.44) | -9.1 (25.34)
  Fatigue, 24 M, FU: number analyzed (Participants) | 70 | 50
  Fatigue, 24 M, FU | -9.1 (23.01) | -11.7 (25.30)
  Financial Difficulties Cycle 4 Day 1: number analyzed (Participants) | 141 | 126
  Financial Difficulties Cycle 4 Day 1 | -4.5 (23.98) | -6.1 (29.93)
  Financial Difficulties, 1 M, FU: number analyzed (Participants) | 136 | 122
  Financial Difficulties, 1 M, FU | -5.9 (26.57) | -5.2 (26.07)
  Financial Difficulties, 3 M, FU: number analyzed (Participants) | 145 | 108
  Financial Difficulties, 3 M, FU | -4.1 (28.30) | -9.0 (29.40)
  Financial Difficulties, 6 M, FU: number analyzed (Participants) | 126 | 98
  Financial Difficulties, 6 M, FU | -5.8 (24.61) | -8.8 (26.89)
  Financial Difficulties, 9 M, FU: number analyzed (Participants) | 114 | 84
  Financial Difficulties, 9 M, FU | -6.1 (27.54) | -8.7 (27.44)
  Financial Difficulties. 12 M, FU: number analyzed (Participants) | 110 | 76
  Financial Difficulties. 12 M, FU | -6.4 (24.93) | -9.6 (28.71)
  Financial Difficulties, 15 M, FU: number analyzed (Participants) | 96 | 62
  Financial Difficulties, 15 M, FU | -8.3 (23.69) | -9.7 (27.91)
  Financial Difficulties, 18 M, FU: number analyzed (Participants) | 90 | 60
  Financial Difficulties, 18 M, FU | -4.1 (24.39) | -12.2 (30.04)
  Financial Difficulties, 21 M, FU,: number analyzed (Participants) | 88 | 51
  Financial Difficulties, 21 M, FU, | -10.6 (22.34) | -11.1 (28.02)
  Financial Difficulties, 24 M, FU: number analyzed (Participants) | 70 | 50
  Financial Difficulties, 24 M, FU | -6.2 (24.93) | -12.0 (27.57)
  Nausea and Vomiting Cycle 4 Day 1: number analyzed (Participants) | 142 | 126
  Nausea and Vomiting Cycle 4 Day 1 | 2.0 (16.06) | 3.7 (18.37)
  Nausea and Vomiting, 1 M, FU: number analyzed (Participants) | 139 | 122
  Nausea and Vomiting, 1 M, FU | 1.0 (14.85) | 0.1 (19.22)
  Nausea and Vomiting, 3 M, FU: number analyzed (Participants) | 145 | 109
  Nausea and Vomiting, 3 M, FU | 0.1 (15.90) | -2.9 (14.49)
  Nausea and Vomiting, 6 M, FU: number analyzed (Participants) | 126 | 99
  Nausea and Vomiting, 6 M, FU | -2.8 (13.12) | -2.5 (14.36)
  Nausea and Vomiting, 9 M, FU: number analyzed (Participants) | 115 | 86
  Nausea and Vomiting, 9 M, FU | -1.3 (13.81) | -1.2 (15.08)
  Nausea and Vomiting. 12 M, FU: number analyzed (Participants) | 110 | 76
  Nausea and Vomiting. 12 M, FU | -2.9 (13.52) | -1.8 (12.35)
  Nausea and Vomiting, 15 M, FU: number analyzed (Participants) | 97 | 62
  Nausea and Vomiting, 15 M, FU | -3.3 (11.45) | -2.7 (11.76)
  Nausea and Vomiting, 18 M, FU: number analyzed (Participants) | 90 | 61
  Nausea and Vomiting, 18 M, FU | -3.3 (12.03) | -2.5 (10.02)
  Nausea and Vomiting, 21 M, FU: number analyzed (Participants) | 88 | 53
  Nausea and Vomiting, 21 M, FU | -4.0 (13.37) | 1.3 (11.72)
  Nausea and Vomiting, 24 M, FU: number analyzed (Participants) | 70 | 50
  Nausea and Vomiting, 24 M, FU | -2.4 (13.69) | -0.3 (11.90)
  Pain Cycle 4 Day 1: number analyzed (Participants) | 142 | 126
  Pain Cycle 4 Day 1 | -3.6 (20.64) | -4.2 (20.43)
  Pain, 1 M, FU: number analyzed (Participants) | 139 | 122
  Pain, 1 M, FU | -2.8 (23.02) | -5.5 (22.31)
  Pain, 3 M, FU: number analyzed (Participants) | 145 | 109
  Pain, 3 M, FU | -3.8 (25.13) | -2.1 (24.44)
  Pain, 6 M, FU: number analyzed (Participants) | 126 | 99
  Pain, 6 M, FU | -5.3 (23.54) | -6.6 (20.59)
  Pain, 9 M, FU: number analyzed (Participants) | 115 | 86
  Pain, 9 M, FU | -4.2 (23.86) | -4.8 (22.12)
  Pain. 12 M, FU: number analyzed (Participants) | 110 | 76
  Pain. 12 M, FU | -3.5 (24.43) | -3.7 (21.01)
  Pain, 15 M, FU: number analyzed (Participants) | 98 | 62
  Pain, 15 M, FU | -2.9 (23.08) | -3.5 (22.00)
  Pain, 18 M, FU: number analyzed (Participants) | 90 | 61
  Pain, 18 M, FU | -3.3 (19.39) | 0.5 (28.05)
  Pain, 21 M, FU: number analyzed (Participants) | 88 | 53
  Pain, 21 M, FU | -5.9 (19.74) | -0.9 (25.82)
  Pain, 24 M, FU: number analyzed (Participants) | 70 | 50
  Pain, 24 M, FU | -1.7 (23.25) | -3.0 (24.67)
  Physical Functioning Cycle 4 Day 1: number analyzed (Participants) | 141 | 124
  Physical Functioning Cycle 4 Day 1 | 1.2 (14.50) | 0.6 (16.81)
  Physical Functioning, 1 M, FU: number analyzed (Participants) | 139 | 122
  Physical Functioning, 1 M, FU | 0.4 (19.52) | -0.7 (21.15)
  Physical Functioning, 3 M, FU: number analyzed (Participants) | 142 | 108
  Physical Functioning, 3 M, FU | 0.9 (18.66) | 0.9 (19.68)
  Physical Functioning, 6 M, FU: number analyzed (Participants) | 124 | 98
  Physical Functioning, 6 M, FU | 3.2 (16.41) | 5.7 (17.01)
  Physical Functioning, 9 M, FU: number analyzed (Participants) | 113 | 83
  Physical Functioning, 9 M, FU | 3.9 (17.30) | 6.2 (17.25)
  Physical Functioning. 12 M, FU: number analyzed (Participants) | 109 | 73
  Physical Functioning. 12 M, FU | 2.4 (17.98) | 3.5 (17.52)
  Physical Functioning, 15 M, FU: number analyzed (Participants) | 96 | 60
  Physical Functioning, 15 M, FU | 3.8 (14.65) | 2.7 (18.46)
  Physical Functioning, 18 M, FU: number analyzed (Participants) | 90 | 60
  Physical Functioning, 18 M, FU | 4.1 (16.65) | 0.1 (22.09)
  Physical Functioning, 21 M, FU: number analyzed (Participants) | 88 | 52
  Physical Functioning, 21 M, FU | 4.7 (17.14) | 2.1 (18.88)
  Physical Functioning, 24 M, FU: number analyzed (Participants) | 69 | 49
  Physical Functioning, 24 M, FU | 5.3 (17.44) | 3.7 (20.57)
  Global Health Status Cycle 4 Day 1: number analyzed (Participants) | 140 | 122
  Global Health Status Cycle 4 Day 1 | 6.4 (23.46) | 6.8 (17.54)
  Global Health Status, 1 M, FU: number analyzed (Participants) | 136 | 119
  Global Health Status, 1 M, FU | 6.5 (24.23) | 6.9 (26.32)
  Global Health Status, 3 M, FU: number analyzed (Participants) | 142 | 105
  Global Health Status, 3 M, FU | 5.0 (21.45) | 12.3 (21.15)
  Global Health Status, 6 M, FU: number analyzed (Participants) | 125 | 97
  Global Health Status, 6 M, FU | 7.5 (21.57) | 13.7 (23.01)
  Global Health Status, 9 M, FU: number analyzed (Participants) | 112 | 83
  Global Health Status, 9 M, FU | 7.6 (23.24) | 11.7 (22.35)
  Global Health Status. 12 M, FU: number analyzed (Participants) | 110 | 74
  Global Health Status. 12 M, FU | 7.6 (23.64) | 12.2 (21.77)
  Global Health Status, 15 M, FU: number analyzed (Participants) | 93 | 61
  Global Health Status, 15 M, FU | 7.6 (20.40) | 12.7 (22.29)
  Global Health Status, 18 M, FU: number analyzed (Participants) | 89 | 60
  Global Health Status, 18 M, FU | 9.2 (23.03) | 10.4 (27.00)
  Global Health Status, 21 M, FU: number analyzed (Participants) | 87 | 53
  Global Health Status, 21 M, FU | 10.8 (20.26) | 12.7 (21.53)
  Global Health Status, 24 M, FU: number analyzed (Participants) | 68 | 48
  Global Health Status, 24 M, FU | 12.1 (24.28) | 12.3 (24.31)
  Role Functioning Cycle 4 Day 1: number analyzed (Participants) | 140 | 124
  Role Functioning Cycle 4 Day 1 | 1.4 (23.27) | 0.1 (24.83)
  Role Functioning, 1 M, FU: number analyzed (Participants) | 138 | 120
  Role Functioning, 1 M, FU | -0.1 (25.83) | -0.7 (27.53)
  Role Functioning, 3 M, FU: number analyzed (Participants) | 141 | 107
  Role Functioning, 3 M, FU | 0.5 (25.19) | 0.9 (28.94)
  Role Functioning, 6 M, FU: number analyzed (Participants) | 124 | 97
  Role Functioning, 6 M, FU | 4.3 (25.49) | 5.5 (26.54)
  Role Functioning, 9 M, FU: number analyzed (Participants) | 113 | 83
  Role Functioning, 9 M, FU | 4.1 (26.21) | 6.2 (25.60)
  Role Functioning. 12 M, FU: number analyzed (Participants) | 109 | 72
  Role Functioning. 12 M, FU | 2.1 (26.46) | 3.9 (24.78)
  Role Functioning, 15 M, FU: number analyzed (Participants) | 96 | 60
  Role Functioning, 15 M, FU | 3.8 (24.84) | 1.9 (25.13)
  Role Functioning, 18 M, FU: number analyzed (Participants) | 90 | 60
  Role Functioning, 18 M, FU | 7.0 (24.09) | -0.0 (28.95)
  Role Functioning, 21 M, FU: number analyzed (Participants) | 88 | 51
  Role Functioning, 21 M, FU | 5.3 (22.82) | 2.6 (26.74)
  Role Functioning, 24 M, FU: number analyzed (Participants) | 69 | 49
  Role Functioning, 24 M, FU | 5.8 (25.54) | 3.7 (30.10)
  Social Functioning Cycle 4 Day 1: number analyzed (Participants) | 142 | 126
  Social Functioning Cycle 4 Day 1 | 3.1 (20.30) | -0.9 (23.50)
  Social Functioning, 1 M, FU: number analyzed (Participants) | 138 | 122
  Social Functioning, 1 M, FU | 0.4 (25.98) | 0.8 (27.93)
  Social Functioning, 3 M, FU: number analyzed (Participants) | 145 | 109
  Social Functioning, 3 M, FU | 0.8 (23.76) | 4.3 (26.29)
  Social Functioning, 6 M, FU: number analyzed (Participants) | 126 | 99
  Social Functioning, 6 M, FU | 3.4 (22.04) | 6.1 (26.24)
  Social Functioning, 9 M, FU: number analyzed (Participants) | 115 | 84
  Social Functioning, 9 M, FU | 2.3 (21.84) | 4.2 (25.46)
  Social Functioning. 12 M, FU: number analyzed (Participants) | 110 | 76
  Social Functioning. 12 M, FU | 3.0 (23.04) | 3.3 (21.95)
  Social Functioning, 15 M, FU: number analyzed (Participants) | 96 | 62
  Social Functioning, 15 M, FU | 6.2 (18.30) | 1.6 (27.61)
  Social Functioning, 18 M, FU: number analyzed (Participants) | 90 | 61
  Social Functioning, 18 M, FU | 6.5 (19.78) | 2.7 (29.69)
  Social Functioning, 21 M, FU: number analyzed (Participants) | 88 | 52
  Social Functioning, 21 M, FU | 6.6 (18.83) | 4.5 (24.72)
  Social Functioning, 24 M, FU: number analyzed (Participants) | 70 | 50
  Social Functioning, 24 M, FU | 7.9 (19.60) | 7.7 (24.56)
  Insomnia Cycle 4 Day 1: number analyzed (Participants) | 138 | 123
  Insomnia Cycle 4 Day 1 | -3.1 (26.07) | -8.7 (26.94)
  Insomnia, 1 M, FU: number analyzed (Participants) | 135 | 120
  Insomnia, 1 M, FU | -5.9 (29.04) | -11.1 (27.78)
  Insomnia, 3 M, FU: number analyzed (Participants) | 139 | 108
  Insomnia, 3 M, FU | -6.2 (29.64) | -13.3 (28.07)
  Insomnia, 6 M, FU: number analyzed (Participants) | 121 | 98
  Insomnia, 6 M, FU | -5.2 (26.18) | -17.0 (25.88)
  Insomnia, 9 M, FU: number analyzed (Participants) | 112 | 81
  Insomnia, 9 M, FU | -3.0 (30.53) | -13.2 (31.04)
  Insomnia. 12 M, FU: number analyzed (Participants) | 106 | 73
  Insomnia. 12 M, FU | -6.9 (25.91) | -10.5 (29.33)
  Insomnia, 15 M, FU: number analyzed (Participants) | 96 | 59
  Insomnia, 15 M, FU | -5.9 (29.02) | -17.5 (26.52)
  Insomnia, 18 M, FU: number analyzed (Participants) | 89 | 59
  Insomnia, 18 M, FU | -7.5 (28.32) | -15.3 (28.58)
  Insomnia, 21 M, FU: number analyzed (Participants) | 86 | 52
  Insomnia, 21 M, FU | -8.5 (25.15) | -10.3 (34.64)
  Insomnia, 24 M, FU: number analyzed (Participants) | 68 | 49
  Insomnia, 24 M, FU | -1.5 (33.30) | -13.6 (35.95)

26. Secondary Outcome: Mean of Health Change Questionnaire (HCQ)
Description: The HCQ consists of a single question in which the participant is asked if he/she has experienced any change in his/her health overall since beginning the study. For HCQ, values from 1 to 9 were assigned to the 9 responses in the HCQ questionnaire, ranging from 1 for 'my health is a great deal better' to 9 for 'my health is a great deal worse' since the beginning of the study. Lower scores represent better conditions.
Time Frame: Screening, Cycle 3 Day 1, and 1 M and every 3 month post last dose up to 24 month.
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183 | 182
Unit on a scale
  Cycle 4 Day 1: number analyzed (Participants) | 139 | 124
  Cycle 4 Day 1 | 2.6 (1.62) | 2.8 (1.59)
  1 M, FU: number analyzed (Participants) | 138 | 121
  1 M, FU | 3.0 (2.05) | 3.2 (2.30)
  3 M, FU: number analyzed (Participants) | 141 | 108
  3 M, FU | 3.0 (2.11) | 2.8 (1.86)
  6 M, FU: number analyzed (Participants) | 124 | 98
  6 M, FU | 2.6 (1.76) | 2.6 (1.82)
  9 M, FU: number analyzed (Participants) | 112 | 85
  9 M, FU | 2.5 (1.78) | 2.4 (1.57)
  12 M, FU: number analyzed (Participants) | 108 | 74
  12 M, FU | 2.5 (1.80) | 2.5 (1.78)
  15 M, FU: number analyzed (Participants) | 96 | 61
  15 M, FU | 2.2 (1.57) | 2.3 (1.68)
  18 M, FU: number analyzed (Participants) | 88 | 58
  18 M, FU | 2.4 (1.67) | 2.7 (2.01)
  21 M, FU: number analyzed (Participants) | 87 | 52
  21 M, FU | 2.3 (1.50) | 2.3 (1.52)
  24 M, FU: number analyzed (Participants) | 69 | 49
  24 M, FU | 2.3 (1.76) | 2.6 (1.89)

27. Secondary Outcome: Mean Area Under the Time-concentration Curve (AUC) Curve Over the Dosing Interval (AUC[0-tau]) of Ofatumumab
Description: Area under the time-concentration curve (AUC) over the dosing interval (AUC[0-tau]) was evaluated. Blood samples were collected from participants who received ofatumumab plus fludarabine and cyclophosphamide predose and 0.5 h after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, predose samples were collected prior to ofatumumab administration at Cycles 2, 3, 5, and 6 (Days 29, 57, 113, and 141).
Time Frame: Cycle 1 Week 1, Cycle 1 Week 2, Cycles 2,3,4,5,6
Population: PK Population: Participants for whom a pharmacokinetic sample was obtained were analyzed, only participants available at the specified time points were analyzed(represented by n=X in the category titles)
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nanogram/mililiter (h*ng/mL)
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183
hour*nanogram/mililiter (h*ng/mL)
  cycle 1, week 1: number analyzed (Participants) | 158
  cycle 1, week 1 | 3554.910 [3224.844 to 3918.759]
  cycle 1, week 2: number analyzed (Participants) | 129
  cycle 1, week 2 | 34109.67 [30042.08 to 38728.00]
  cycle 2: number analyzed (Participants) | 147
  cycle 2 | 67069.79 [59485.45 to 75621.13]
  cycle 3: number analyzed (Participants) | 129
  cycle 3 | 84620.05 [76209.86 to 93958.35]
  cycle 4: number analyzed (Participants) | 107
  cycle 4 | 89091.35 [78326.34 to 101335.9]
  cycle 5: number analyzed (Participants) | 97
  cycle 5 | 96829.23 [84488.81 to 110972.1]
  cycle 6: number analyzed (Participants) | 91
  cycle 6 | 104798.0 [90904.74 to 120814.6]

28. Secondary Outcome: Maximum Concentration (Cmax) and Observed Drug Concentration Prior to the Next Dose (Ctrough) of Ofatumumab
Description: Blood samples were collected to assess the plasma concentration of ofatumumab.Cmax and Ctrough were determined. Blood samples were collected from participants who received ofatumumab plus fludarabine and cyclophosphamide predose and 0.5 h after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, predose samples were collected prior to ofatumumab administration at Cycles 2, 3, 5, and 6 (Days 29, 57, 113, and 141).
Time Frame: Cycle 1 Week 1, Cycle 1 Week 2, Cycles 2,3,4,5
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183
Micrograms per milliliter
  Cmax cycle 1, week 1: number analyzed (Participants) | 154
  Cmax cycle 1, week 1 | 61.355 [55.444 to 67.897]
  Cmax cycle 1, week 2: number analyzed (Participants) | 159
  Cmax cycle 1, week 2 | 241.192 [210.492 to 276.369]
  Cmax cycle 4: number analyzed (Participants) | 140
  Cmax cycle 4 | 312.745 [287.708 to 339.961]
  Ctrough cycle 1, week 1: number analyzed (Participants) | 167
  Ctrough cycle 1, week 1 | 3.551 [2.417 to 5.217]
  Ctrough cycle 1, week 2: number analyzed (Participants) | 165
  Ctrough cycle 1, week 2 | 9.496 [6.565 to 13.736]
  Ctrough cycle 2: number analyzed (Participants) | 162
  Ctrough cycle 2 | 24.281 [17.953 to 32.840]
  Ctrough cycle 3: number analyzed (Participants) | 150
  Ctrough cycle 3 | 25.632 [18.884 to 34.791]
  Ctrough cycle 4: number analyzed (Participants) | 130
  Ctrough cycle 4 | 58.640 [44.465 to 77.333]
  Ctrough cycle 5: number analyzed (Participants) | 113
  Ctrough cycle 5 | 70.398 [55.257 to 89.686]

29. Secondary Outcome: Time of Occurrence of Cmax (Tmax) of Ofatumumab
Description: Blood samples were collected from participants who received ofatumumab plus fludarabine and cyclophosphamide predose and 0.5 h after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4.
Time Frame: Cycle 1 Week 1, Cycle 1 Week 2, Cycle 4
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects
Number analyzed (Participants) | 183
Hour
  cycle 1, week 1: number analyzed (Participants) | 154
  cycle 1, week 1 | 6.106 [5.789 to 6.442]
  cycle 1, week 2: number analyzed (Participants) | 159
  cycle 1, week 2 | 5.004 [4.896 to 5.114]
  cycle 4: number analyzed (Participants) | 140
  cycle 4 | 4.878 [4.661 to 5.105]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 5 years.
Description: Analysis was done in the safety Population included subjects who received at least one dose of a study drug. This population was used for all safety measurements. In the analyses, subjects were grouped based on the treatment they receive regardless of how they are randomized.
Arm/Group | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects | Fludarabine + Cyclophosphamide_ ITT Subjects
All-Cause Mortality (participants affected / at risk) | 40/181 | 42/178
Serious Adverse Events (participants affected / at risk) | 108/181 | 86/178
Other Adverse Events (participants affected / at risk) | 149/181 | 123/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects (N=181) | Fludarabine + Cyclophosphamide_ ITT Subjects (N=178)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 11 | 12
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 15
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 17 | 14
Pancytopenia (Blood and lymphatic system disorders) | 5 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 10
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 3
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 4
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Epidermolysis (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 2
Hyperthermia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 9 | 5
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis salmonella (Infections and infestations) | 2 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 1
Hepatitis B reactivation (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 2
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 2
Neutropenic infection (Infections and infestations) | 0 | 2
Neutropenic sepsis (Infections and infestations) | 4 | 5
Oral candidiasis (Infections and infestations) | 0 | 2
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 28 | 29
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Salmonella sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 8
Septic shock (Infections and infestations) | 1 | 3
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Systemic mycosis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 6 | 6
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Starvation (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 2
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 1
Haemorrhagic vasculitis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Fludarabine + Cyclophosphamide_ ITT Subjects (N=181) | Fludarabine + Cyclophosphamide_ ITT Subjects (N=178)
Anaemia (Blood and lymphatic system disorders) | 24 | 38
Leukopenia (Blood and lymphatic system disorders) | 27 | 10
Neutropenia (Blood and lymphatic system disorders) | 93 | 62
Thrombocytopenia (Blood and lymphatic system disorders) | 38 | 55
Constipation (Gastrointestinal disorders) | 8 | 11
Diarrhoea (Gastrointestinal disorders) | 14 | 19
Nausea (Gastrointestinal disorders) | 45 | 36
Vomiting (Gastrointestinal disorders) | 19 | 22
Asthenia (General disorders) | 13 | 16
Chills (General disorders) | 14 | 3
Fatigue (General disorders) | 15 | 11
Pyrexia (General disorders) | 26 | 15
Upper respiratory tract infection (Infections and infestations) | 13 | 8
Platelet count decreased (Investigations) | 12 | 5
Decreased appetite (Metabolism and nutrition disorders) | 13 | 8
Headache (Nervous system disorders) | 15 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 2
Rash (Skin and subcutaneous tissue disorders) | 23 | 8
Hypotension (Vascular disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.